CLINICAL TRIAL: NCT04070703
Title: Efficacy of Adapted Tai Ji Quan to Slow Cognitive Decline in Older Adults
Brief Title: Tai Ji Quan and Cognitive Function in Older Adults With Mild Cognitive Impairment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AG059546
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognitive function; mild cognitive impairment; Tai Ji Quan
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitively enhanced Tai Ji Quan (Experimental): Participants in this arm will exercise a series of Tai Ji Quan-based movements with configurations that are specifically designed for older adults to improve cognitive function, dual-task ability, strength/balance, and mobility.
  Interventions: Behavioral: The Go for Exercise & Healthy Aging Project
- Standard Tai Ji Quan (Active Comparator): Serving as an active comparison arm, participants in this intervention will exercise a series of Tai Ji Quan-based movements that are specifically designed for older adults to improve strength/balance, cognitive function, and mobility.
  Interventions: Behavioral: The Go for Exercise & Healthy Aging Project
- Stretching (Sham Comparator): Serving as a control arm, participants in this intervention will engage in a series of light exercise activities consisting of breathing, stretching, and body relaxation.
  Interventions: Behavioral: The Go for Exercise & Healthy Aging Project

INTERVENTIONS:
Behavioral: The Go for Exercise & Healthy Aging Project — Exercise and Cognition

SUMMARY:
To determine the efficacy of a cognitively enhanced exercise intervention - Tai Ji Quan: Moving to Maintain Brain Health in improving global cognitive function and dual-task ability in older adults with mild cognitive impairment.

DETAILED DESCRIPTION:
The primary aim of the study is to determine the efficacy of a cognitively enhanced exercise intervention - Tai Ji Quan: Moving to Maintain Brain Health, relative to a standard Tai Ji Quan intervention and an exercise stretching control, in improving global cognitive function and dual-task ability among community-dwelling older adults with amnestic mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* complaint of memory loss
* clinical dementia rating (CDR) scale score ≤0.5
* having normal general cognitive function screened, with MMSE ≥24
* capable of exercising safely, as determined by a healthcare provider
* willingness to be randomly assigned to an intervention condition and complete the 24-week intervention and 6-month follow-up

Exclusion Criteria:

* having medical conditions likely to compromise survival, such as metastatic cancer, or render a participant unable to engage in physical activity, such as severe cardiac failure
* participating in any type of Tai Ji Quan or daily and/or structured vigorous physical activity (i.e., brisk walking for exercise 30 minutes or longer at a time, or engaging in muscle-strengthening activities, e.g., weight lifting on 3 or more days per week 3 months prior to the study)

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 318 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Fuzhong Li, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
The individual level data in this study will not be shared with others for reasons of confidentiality. However, a dataset with identifiable private information removed may be made available to other researchers.

REFERENCES:
- [Background] Li F, Harmer P, Eckstrom E, Fitzgerald K, Winters-Stone K. Clinical Effectiveness of Cognitively Enhanced Tai Ji Quan Training on Global Cognition and Dual-Task Performance During Walking in Older Adults With Mild Cognitive Impairment or Self-Reported Memory Concerns : A Randomized Controlled Trial. Ann Intern Med. 2023 Nov;176(11):1498-1507. doi: 10.7326/M23-1603. Epub 2023 Oct 31. PMID 37903365
- [Derived] Li F, Harmer P, Eckstrom E, Winters-Stone K. Physical Activity Engagement After Tai Ji Quan Intervention Among Older Adults With Mild Cognitive Impairment or Memory Concerns: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Dec 2;7(12):e2450457. doi: 10.1001/jamanetworkopen.2024.50457. PMID 39688866
- [Derived] Li F, Harmer P, Fitzgerald K, Winters-Stone K. A cognitively enhanced online Tai Ji Quan training intervention for community-dwelling older adults with mild cognitive impairment: A feasibility trial. BMC Geriatr. 2022 Jan 25;22(1):76. doi: 10.1186/s12877-021-02747-0. PMID 35078407
- See also: published article — https://pubmed.ncbi.nlm.nih.gov/37903365/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Started | 105 | 107 | 106
Completed | 102 | 103 | 99
Not Completed | 3 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching | Total
Number analyzed (Participants) | 105 | 107 | 106 | 318
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 105 | 107 | 106 | 318
Age, Continuous [Mean (Standard Deviation); unit: years] — Age measured in year
  years | 76 (5) | 76 (5) | 76 (5) | 76 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 66 | 71 | 212
  Male | 30 | 41 | 35 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 4 | 14
  Not Hispanic or Latino | 96 | 90 | 89 | 275
  Unknown or Not Reported | 5 | 11 | 13 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 4 | 7
  White | 96 | 90 | 89 | 275
  More than one race | 6 | 13 | 9 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Participants were recruited from 81 cities/towns across 25 states in the U.S. The detailed number from each state is not shown.
  Participants
    United States | 105 | 107 | 106 | 318

OUTCOME MEASURES:

1. Primary Outcome: Montreal Cognitive Assessment
Description: The Montreal Cognitive Assessment scale measures change in global cognitive function from baseline to 6 months. The scale scores range from 0 to 30 points, with higher scores indicating better cognitive functioning.
Time Frame: baseline, 6 months
Population: The primary outcome data were analyzed via a Group by Time mixed-effects model with repeated measures on the second factor (i.e., outcome measures assessed at baseline and 6 months. In the presence of a Group by Time interaction effect, pre-specified follow-up pair-wise comparisons were performed to determine between-group differences.
Measure: Mean (Standard Error); unit: points
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
points
  Baseline | 25.2 (0.2) | 25.3 (0.2) | 25.3 (0.2)
  Int Termination | 28.4 (.2) | 27 (.2) | 25.6 (.2)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority — The co-primary outcome data were analyzed via a Group by Time mixed-effects model with repeated measures on the second factor (i.e., outcome measures assessed at baseline and 6 months. In the presence of a Group by Time interaction effect, pre-specified follow-up pair-wise comparisons were performed to determine between-group differences; p = 0.0125, Mixed Models Analysis; Mean Difference (Final Values) = 2.8, 98.75% CI 2-sided [2.1 to 3.6]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p = .0125, Mixed Models Analysis; Mean Difference (Final Values) = 1.5, 98.75% CI 2-sided [.07 to 2.2]

2. Primary Outcome: Gait Performance Under a Dual-task Condition
Description: Assessing change in dual-task ability (measured in seconds) from baseline to 6 months. Change will be assessed via an Instrumental Timed Up&Go (iTUG) gait performance (APDM, Inc.) in which the participant is asked to stand up from a chair, walk a 6-m walkway at normal pace (3 m toward a line, turn, and 3 m toward the chair), turn around, and sit down on the chair, with no cognitive task (single-task walking). The participant is then asked to perform the same procedure with a concurrent cognitive task (counting backward by 3s, starting with an odd number, e.g., 81).12 The total walking duration (in seconds) during both 6-meter walks, at normal pace, will be recorded. Lower duration indicates a better outcome.
Time Frame: baseline, 6 months
Population: The co-primary outcome data were analyzed via a Group by Time mixed-effects model with repeated measures on the second factor (i.e., outcome measures assessed at baseline and 6 months. In the presence of a Group by Time interaction effect, pre-specified follow-up pair-wise comparisons were performed to determine between-group differences.
Measure: Mean (Standard Error); unit: second
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
second
  baseline | 36.3 (2.3) | 36.3 (2.3) | 36.3 (2.4)
  6 months | 15.5 (1.6) | 25.2 (1.5) | 37.5 (1.6)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p = .0125, Mixed Models Analysis; Mean Difference (Final Values) = 9.9, 98.75% CI 2-sided [2.8 to 16.6]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p = .0125, Mixed Models Analysis; Mean Difference (Final Values) = 22, 98.75% CI 2-sided [12.6 to 31.2]

3. Secondary Outcome: Clinical Dementia Rating Scale
Description: The Clinical Dementia Rating Scale measures change in cognitive decline from baseline to 6 months. The scale measures six domains of cognitive and functional performance. Scores range from 0 to 3 points in each domain, with a score of 0 indicating no impairment, while a score of 3 signifying severe impairment. Scores from all domains have been averaged to compute the total score reported. In this trial, lower scores indicate less severity in cognitive decline (i.e., improvement from intervention).
Time Frame: baseline, 6 months
Population: Analysis of variance examining difference between groups
Measure: Mean (Standard Error); unit: points
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
points
  baseline | 1.0 (.1) | 1.1 (.1) | 1.1 (.1)
  6 months | .3 (.1) | .6 (.1) | .9 (.1)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-.5 to -.1]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p = .05, Mixed Models Analysis; Mean Difference (Final Values) = -.6, 95% CI 2-sided [-.7 to -.3]

4. Secondary Outcome: Domain-specific Cognitive Test - Trail Making - B
Description: Change in domain-specific cognitive function - executive function (measured in seconds) from baseline to 24 weeks. Trail Making Test assesses attention and executive function. In this test, the participant connects numbers and letters in an alternating progressive sequence, 1 to A, 2 to B, 3 to C, and so on. For parts A and B, scoring is expressed in terms of the time (in seconds) to completion. Lower scores indicate higher executive functioning.
Time Frame: baseline, 6 months
Population: Analysis of variance examining difference between groups.
Measure: Mean (Standard Error); unit: second
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
second
  baseline | 98.7 (1.6) | 98.4 (1.5) | 98 (1.6)
  6 months | 72.4 (2.0) | 86.2 (2.0) | 94.2 (2.1)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p = .05, Mixed Models Analysis; Mean Difference (Final Values) = -14.1, 95% CI 2-sided [-20 to -8]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p = .05, Mixed Models Analysis; Mean Difference (Final Values) = -22, 95% CI 2-sided [-28 to -16]

5. Secondary Outcome: 4-Stage Balance Test
Description: The 4-Stage Balance Test measures change, from baseline to 6 months, in standing four positions balance. Participants attempt to hold four progressively challenging standing positions. The test ends if a position cannot be held for 10 seconds. The number of positions successfully completed is recorded and awarded one point (0-4), with higher score values indicating better balance.
Time Frame: baseline, 6 months
Population: analysis of variance examining differences between groups.
Measure: Mean (Standard Error); unit: points
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
points
  baseline | 2.6 (.1) | 2.6 (.1) | 2.6 (.1)
  6 months | 3.4 (.1) | 3.5 (.1) | 2.6 (.1)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = .1, 95% CI 2-sided [-.4 to .1]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = .8, 95% CI 2-sided [.4 to 1.2]

6. Secondary Outcome: Backward Digit Span
Description: The Backward Digit Span test assesses memory. The participant is verbally presented with a series of digits (e.g., 6, 2, 9, 7) at a rate of one digit per second and is required to repeat them verbatim. If the participant succeeds, he/she is given a longer list (e.g., 5, 3, 8, 1, 6). The number of digits increases by one until the participant consecutively fails two trials of the same digit span length. The length of the longest list a person can remember is that person's digit span. In this test, the participant is required to repeat the digits in reverse. The participant receives 1 point for each correct answer. The Backward Digit Span test scores range from 0 to 32, with higher scores indicating better memory.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
points
  baseline | 8.3 (.2) | 8.4 (.2) | 8.4 (.2)
  6 months | 10.4 (.2) | 9.4 (.2) | 8.3 (.2)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [.5 to 1.6]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [1.6 to 2.7]

7. Secondary Outcome: Verbal Fluency Test
Description: The Verbal Fluency Test assesses verbal fluency and executive function of cognitive function. The participant is asked to generate the names of as many animals as possible in 60 seconds. High scores (i.e., more animals names generated) in this measure indicate better performance (i.e., better verbal fluency and executive function).
Time Frame: baseline, 6 months
Measure: Mean (Standard Error); unit: number of animals
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
number of animals
  baseline | 14 (.2) | 14 (.2) | 14 (.2)
  6 months | 19 (.3) | 19 (.3) | 15 (.3)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = .9, 95% CI 2-sided [-.4 to 2.1]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 4.4, 95% CI 2-sided [3.1 to 5]

8. Secondary Outcome: Timed up and go
Description: The Timed up and go (TUG) measure is recorded in seconds (the time taken by an individual to stand up from a standard armless chair, walk a distance of 3 meters, turn, walk back to the chair, and sit down). Lower scores indicate better performance.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
seconds
  baseline | 12.6 (.2) | 12.7 (.2) | 12.5 (.3)
  6 months | 10.8 (.2) | 10.6 (.2) | 12.6 (.3)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = .3, 95% CI 2-sided [-.3 to .7]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.4 to -1.4]

9. Secondary Outcome: 30-Second Chair Stands Test
Description: The 30-Second Chair Stands Test is used to measure change from baseline to 6 months in physical performance. The Test involves repeatedly standing up from and sitting down in a chair as many times as possible within 30 seconds, with high (count) scores indicating better performance (i.e., leg strength).
Time Frame: baseline, 6 months
Measure: Mean (Standard Error); unit: chair stands
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
chair stands
  baseline | 11 (.2) | 11 (.2) | 11 (.3)
  6 months | 13 (.4) | 13 (.4) | 11 (.4)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = -.4, 95% CI 2-sided [-1.4 to .4]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [.8 to 2.3]

10. Secondary Outcome: Forward Digit Span Test
Description: The Forward Digit Span test measures attention/concentration (in points) with high scores indicating better attention. The participant is verbally presented with a series of digits (e.g., 6, 2, 9, 7) at a rate of one digit per second and is required to repeat them verbatim. If the participant succeeds, he/she is given a longer list (e.g., 5, 3, 8, 1, 6). The number of digits increases by one until the participant consecutively fails two trials of the same digit span length. The length of the longest list a person can remember is that person's digit span.
Time Frame: baseline, 6 months
Population: analysis of variance was conducted examining differences between groups
Measure: Mean (Standard Error); unit: point
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
point
  baseline | 12.8 (.1) | 10.6 (.1) | 10.7 (.1)
  6 months | 10.4 (.2) | 9.4 (.2) | 8.3 (.2)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = .5, 95% CI 2-sided [-.1 to 1.1]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [1.6 to 2.8]

11. Other Pre Specified Outcome: Sleep Quality - Pittsburgh Sleep Quality Index (PSQI)
Description: Change in sleep quality from baseline to 24 weeks. The Pittsburgh Sleep Quality Index (PSQI) includes seven indices: subjective quality, latency (i.e., time needed to fall asleep), duration (i.e., number of hours of actual sleep per night), efficiency (i.e., total sleep time divided by time in bed, converted to a score of 0-3), sleep disturbances (e.g., waking up in the middle of the night and the like), use of sleeping medication, and daytime dysfunction (e.g., having difficulty staying awake during the day). Each of the component scores ranges from 0 to 3, with the PSQI global score ranging from 0 to 21 points, with higher scores indicating poorer sleep quality.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
points
  baseline | 8.2 (.3) | 8.3 (.3) | 8.1 (.3)
  6 months | 5.2 (.3) | 5.2 (.3) | 7.3 (.3)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = .1, 95% CI 2-sided [-.7 to .8]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-3.1 to -1.3]

12. Other Pre Specified Outcome: Depression - Geriatric Depression Scale (GDS)
Description: Change in depression from baseline to 24 weeks. The Geriatric Depression Scale (GDS) score ranges from 0 to 15 with higher scores indicated increased depression symptoms and scores higher than 5 indicative of depression.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
points
  baseline | 3.5 (.3) | 3.4 (.3) | 3.4 (.3)
  6 months | 1.6 (.2) | 1.2 (.2) | 2.5 (.2)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = .5, 95% CI 2-sided [-.3 to 1.2]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = -1, 95% CI 2-sided [-1.8 to -.2]

13. Other Pre Specified Outcome: Activity and Movement Confidence Scales
Description: The Activity and Movement Confidence Scales measure a person's movement confidence. In this study it assesses change in activity and movement confidence from baseline to 24 weeks. The total score ranges from 0 to 100 with higher scores indicating higher confidence.
Time Frame: baseline, 6 months
Population: Analysis of variance was conducted to examine differences between groups
Measure: Mean (Standard Deviation); unit: point
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
point
  baseline | 82 (1.3) | 82.6 (1.3) | 81.6 (1.3)
  6 months | 89.5 (1.3) | 88.3 (1.3) | 83.1 (1.3)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-.4 to 2]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [3.1 to 7.9]

14. Other Pre Specified Outcome: Quality of Life - EuroQol.
Description: The Quality of Life - EuroQol. scale assesses quality of life. Change in quality of life from baseline to 24 weeks. The EQ-5D-3L version will be used that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The scores of EQ-5D-3L will be averaged to generate a single utility value ranging from 1.00 for the "best health" state to -0.594 for the "worst health" state, where a score of 0 is indicative of death, and scores less than 0 are considered as "worse than death." Participants who die during the trial period will be registered as 0 in utility terms for the assessment period from when the death occurred.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
points
  baseline | .76 (.01) | .77 (.01) | .77 (.01)
  6 months | .90 (.01) | .90 (.01) | .76 (.01)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = -.0, 95% CI 2-sided [-.04 to .03]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = .07, 95% CI 2-sided [.03 to .11]

15. Other Pre Specified Outcome: International Physical Activity Questionnaire (IPAQ)
Description: The International Physical Activity Questionnaire (IPAQ) measures the level of moderate and vigorous physical activity (MVPA) (measured in minutes) with high scores indicating high level of physical activity. This measure asks participants to report how often (measured in days) and how much time (in minutes) over the previous week they participated in physical activity or exercise of any moderate (ex. gardening, cleaning, etc.) or vigorous (ex. heavy lifting, jogging/running or fast bicycling, etc.) intensity that lasted at least 10 minutes at a time. The activities to be asked during the post-intervention follow-up (at 6 months) will not include the time spent in attending the assigned exercise programs in the study. Total weekly duration of MVPA, measured in minutes, are calculated by multiplying frequency and duration (vigorous activity weighted by 2) to form a total weighted amount of MVPA min/week.
Time Frame: baseline and 6 months
Population: Analysis of variance was conducted to examine differences between groups.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
minutes
  baseline | 146 (12) | 145 (12) | 145.8 (12.3)
  6 months | 273 (12.5) | 267.9 (12) | 147.6 (12.6)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 4, 95% CI 2-sided [-2 to 6]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 125.5, 95% CI 2-sided [84 to 166]

16. Other Pre Specified Outcome: Everyday Cognition Scale
Description: The Everyday Cognition Scale measures change from baseline to 6 months in everyday cognitive function. Sub scale scores will be averaged to create a total score. Total scores range 1 to 4, with higher scores indicating better everyday cognitive function.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
Number analyzed (Participants) | 105 | 107 | 106
points
  baseline | 2 (.04) | 2 (.04) | 2.1 (.04)
  6 months | 1.2 (.1) | 1.4 (.1) | 1.8 (.1)
Statistical Analysis 1: Comparison: Cognitively Enhanced Tai Ji Quan vs Standard Tai Ji Quan; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = -.2, 95% CI 2-sided [-.3 to -.1]
Statistical Analysis 2: Comparison: Cognitively Enhanced Tai Ji Quan vs Stretching; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = -.5, 95% CI 2-sided [-.7 to -.4]

ADVERSE EVENTS:
Time Frame: Events were observed and documented during the 6-month active intervention period.
Description: Data reported in this record is consistent with the definitions described at clinicaltrials.gov
Arm/Group | Cognitively Enhanced Tai Ji Quan | Standard Tai Ji Quan | Stretching
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/107 | 0/106
Serious Adverse Events (participants affected / at risk) | 3/105 | 2/107 | 2/106
Other Adverse Events (participants affected / at risk) | 10/105 | 10/107 | 11/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitively Enhanced Tai Ji Quan (N=105) | Standard Tai Ji Quan (N=107) | Stretching (N=106)
Serious event (General disorders) | 3 (3) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitively Enhanced Tai Ji Quan (N=105) | Standard Tai Ji Quan (N=107) | Stretching (N=106)
Other events (Musculoskeletal and connective tissue disorders) | 10 (10) | 10 (10) | 11 (11) — events that required no or medical treatment and were non-life threatening (e.g., lower back pain, ankle/muscle soreness or pain without needing medical attention).

LIMITATIONS AND CAVEATS:
Limitations of the trial included (a) the lack of a nonexercise control group and (b) participants who were predominately White and well educated which limits the generalizability of these reports.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT04070703/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT04070703/SAP_001.pdf